CLINICAL TRIAL: NCT04924907
Title: Lifestyles, Arterial Aging and Its Relationship With the Intestinal Microbiota (MIVAS III Study)
Brief Title: Lifestyles, Arterial Aging and Intestinal Microbiota (MIVAS III Study)
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Castilla-León Health Service (Other)
Responsible Party: Sponsor
Other Study IDs: PI20/00321; GRS 2148/B/2020 (Other Grant/Funding Number: Gerencia Regional de Salud de Castilla y Leon); GRS 2263/B/2020 (Other Grant/Funding Number: Gerencia Regional de Salud de Castilla y Leon)
Record Dates: First submitted 2021-04-25; First posted 2021-06-14 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2023-12

CONDITIONS: Arterial Stiffness; Dysbiosis
Keywords: Lifestyles; pulse wave velocity; intestinal microbiota; multicentric study
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dysbiosis microbiota: microbiota with proinflammatory pattern or dysbiosis
- Normal microbiota: microbiota with antiinflammatory pattern or normal

SUMMARY:
This is an observational cross-sectional study whose objective is to analyse associations between the intestinal and salivate microbiota with lifestyles (eating patterns, physical activity, tobacco and alcohol consumption), arterial aging and cognitive function. It will take place in five different research units located in Spain

DETAILED DESCRIPTION:
Aim: To analyze the association of lifestyles (eating patterns, physical activity, tobacco and alcohol consumption) with the intestinal and salivate microbiota and its relationship with arterial aging and cognitive function in subjects without cardiovascular disease in Spain and Portugal. In addition, the mediating role of the intestinal microbiota in the relationship of lifestyles with arterial aging and cognitive function will be analyzed.

Design: A cross-sectional study with a case-control analysis, to analyze the association of microbiota patterns with arterial ageing. Setting: the study will develop the research network in health prevention and promotion (Rediapp) and in the Iberian network on arterial structure and the Cancer Research Center of Salamanca. Study population: 1000 subjects aged 45 to 74 years without cardiovascular disease, will be selected.

Variables: Demographic, anthropometric and habits (tobacco and alcohol). A dietary pattern through a frequency consumption questionnaire (FFQ), the software of the EVIDENT III and the Mediterranean Diet adherence questionnaire. Physical activity: International Physical Activity Questionnaire (IPAQ), Marshall Questionnaire and Accelerometer, Actigraph. Body composition (Inbody 230 impedance meter). Arterial aging: Medium intimate carotid thickness (Sonosite Micromax); Analysis (PWA) and pulse wave velocity (cf-PWV), (Sphygmocor System). Cardio Ankle Vascular Index (CAVI), ba-PWV and ankle-brachial index (Vasera VS-2000®). With Ambulatory Pulse Wave Analysis (Microsoft®), the PAIx and CAIx and the heart rate variability will be measured. The vascular damage in the retina, heart, kidney, brain and cardiovascular risk will be measured. Intestinal microbiota with the OMNIgene GUT kit (OMR -200) and analysis of the 16S rRNA microbiome profile by massive sequentiation. (Lifestyles, arterial aging, neurocognition, microbiota)

ELIGIBILITY:
Inclusion Criteria:

* People aged 45 to74 years who agree to participate in the study and who not meet any of the exclusion criteria

Exclusion Criteria:

* Participants with a personal history of cardiovascular disease (ischaemic heart disease or stroke, peripheral arterial disease or Heart Failure)
* Participants with a BMI> 40 kg / m2
* Participants diagnosed renal failure in terminal stages (GFR <30 ml / min);
* Chronic intestinal inflammatory disease or acute inflammatory process in the past 3 months
* Oncology disease diagnosed in the last 5 years or with active treatment
* Participants who are in a terminal condition
* Consumption of antibiotics last 15 days

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged 45 to 74 years without cardiovascular disease
Sampling Method: Probability Sample
Enrollment: 1015 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Pulse Wave Velocity | 1 year
  Measurement by SphygmoCor System (meters/seg)

SECONDARY OUTCOMES:
Physical Activity | 1 year
  Measurement by the International Physical Activity Questionnaire (IPAQ) (min/day)
Eating habits | 1 year
  Measurement by Food Frequency Questionnaire (FFQ) (kcal/day)
Smoking | 1 year
  Measurement by a questionnaire of four questions adapted from the WHO MONICA study (Smoking status and cigarettes frequency)
Drinking habits | 1 year
  Measurement by a frequency alcohol questionnaire (units/day)
Body composition | 1 year
  Measurement by Inbody 230 device (kg)
Carotid intima-media thickness (IMT) | 1 year
  Measurement by Sonosite Micromax Ultrasound (mm)
Cardio Ankle Vascular Index (CAVI) | 1 year
  Measurement by Vasera device 2000 (not units)
Cognitive evaluation | 1 year
  Measurement by Montreal Cognitive Assessment (MOCA) (points). Range: 0-30 points. A score of 26 points or above is considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Garcia-Ortiz, Study Director — Primary Care Research Unit of Salamanca (APISAL); Rita Salvado-Martins, Principal Investigator — Primary Care Research Unit; Pedro Guimaraes-Cunha, Study Director — Life and Health Sciences Research Institute in Minho University
Locations (2):
- Spain (2):
  - Primary Care Research Unit (APISAL), Salamanca
  - Primary Care Research Unit-Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lugones-Sanchez C, Santos-Minguez S, Salvado R, Gonzalez-Sanchez S, Tamayo-Morales O, Hoya-Gonzalez A, Ramirez-Manent JI, Magallon-Botaya R, Quesada-Rico JA, Garcia-Cubillas MD, Rodriguez-Sanchez E, Gomez-Marcos MA, Benito-Sanchez R, Mira A, Hernandez-Rivas JM, Garcia-Ortiz L; MIVAS III Researchers Group. Lifestyles, arterial aging, and its relationship with the intestinal and oral microbiota (MIVAS III study): a research protocol for a cross-sectional multicenter study. Front Public Health. 2023 Jun 29;11:1164453. doi: 10.3389/fpubh.2023.1164453. eCollection 2023. PMID 37457284